CLINICAL TRIAL: NCT04291443
Title: Detection of Orthodontically Induced Inflammatory Root Resorption From Gingival Crevicular Fluid by Proteomics Analysis: Split Mouth, Randomized Clinical Trial
Brief Title: Proteomics and Orthodontic Root Resorption
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Baghdad (Other)
Responsible Party: Principal Investigator, Harraa S. Mohammed-Salih, PhD student, University of Baghdad
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: 023418
Record Dates: First submitted 2020-02-25; First posted 2020-03-02 (Actual); Last update posted 2020-03-02 (Actual); Status verified 2020-02

CONDITIONS: Root Resorption; Orthodontic Appliance Complication; Orthodontic Pathological Resorption of External Root; Gingival Diseases; Tooth Plaque; Tooth Diseases
Keywords: Proteomic; Orthodontic Root Resorption; Gingival Crevicular Fluid
MeSH Terms: conditions — Root Resorption; Gingival Diseases; Dental Plaque; Tooth Diseases

STUDY DESIGN:
Intervention Model Description: Adult orthodontic patients
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The GCF measures were coded by a clinician who bonded the appliance using patient ID number and the side of the arch (either right or left sides) to which orthodontic force (either heavy or light force) was allocated blindly for the investigator and outcomes assessor because the clinician could know the type of force from the shape of archwires. The surgeon who extract the teeth was also blinded. The extracted premolars were coded to be masked to the investigator who measured the root resorption areas. All outcome assessors of proteomic analysis as well as the statistician was blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Upper First Premolar One Side (Experimental): Heavy force (225 g)
  Interventions: Procedure: Heavy Force (225g)
- Upper First Premolar Other Side (Experimental): Light Force (25 g)
  Interventions: Procedure: Light Force (25g)

INTERVENTIONS:
Procedure: Heavy Force (225g) — Orthodontic Force
  Arms: Upper First Premolar One Side
Procedure: Light Force (25g) — Orthodontic Force
  Arms: Upper First Premolar Other Side

SUMMARY:
The majority of previous studies for early detection of Orthodontically Induced Inflammatory Root Resorption (OIIRR) were conducted to assess individual biomarkers which are representative of single biological pathway. To our Knowledge, no studies have been employed Gingival crevicular fluid (GCF) proteomic analysis to identify potential biomarkers for OIIRR. Therefore; the aim of this study is to use the advantage of testing a package of biomarkers via doing proteomic analysis of GCF which could help in making a more precise personalize diagnosis and treatments, thereby providing orthodontists additional information that cannot be deduced from clinical parameters.

DETAILED DESCRIPTION:
Orthodontic patients with age range (18-years) indicated for bilateral maxillary first premolars extraction as part of their orthodontic treatment using specific fixed orthodontic appliance design with moderate anchorage were recruited for this study. Both of these premolars were allocated randomly to a heavy ( 225g) and light (25g) force in a split mouth design with a 1:1 allocation ratio. (GCF) was collected from the gingival sulcus of these teeth before extraction at six time intervals which are baseline, 1 hour, 1 day, 1 week , 2 weeks, 3 weeks and 4 weeks. Plaque and Gingival Indices were recorded for those patients at each timeline. Premolars will be extracted after 4weeks to be examined by stereomicroscopy for surface area evaluation of root resorption. Proteomic analysis will be carried out on the GCF sample. The proteomic analysis of the collected GCF will be obtained by using matrix-assisted laser desorption ionization/ time-of-flight mass spectrometry (MALDI-TOF/MS). MS spectra will be used to search human protein sequence data bases for protein identification and the development of "Protein Print" specific for these biological conditions.

ELIGIBILITY:
Inclusion Criteria:

* Orthodontic patients indicated for extraction of bilateral upper first premolars,
* General healthy fit,
* Good oral hygiene with periodontal health maintenance (Plaque Index and Gingival Index ≤1),
* Lack of radiographic signs of idiopathic resorption,
* Radiographically both experimental teeth have two roots with approximately equal length and shape,
* The position of experimental teeth within the arch with no rotation.

Exclusion Criteria:

* Patients with impaction except impacted third molars for referral to do CBCT,
* Smokers,
* Patients on anti-inflammatory drugs at least three months before and during the study,
* History of oral habit,
* Previous orthodontic treatment,
* History of dental trauma,
* Previous dental treatment of the experimental teeth,
* Patient with heavy occlusion,
* Pathological lesion in the upper arch.

Ages: 18 Years to 32 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
Biomarkers of Orthodontic Root Resorption | Baseline, 1hour, 1day, 7days, 14days, 21days and 28days
  To monitor change in profiling of GCF proteins associated with orthodontically induced root resorption during 4 weeks after orthodontic force application

SECONDARY OUTCOMES:
GCF Flow Rate and Orthodontic Force | Baseline, 1hour, 1day, 7days, 14days, 21days and 28days
  To determine the impact of different orthodontic force magnitudes on GCF flow rate
Root Resorption Surface Area | After 28 days of force application.
  To estimate the amount of resorption area in different force groups.
Protein concentration in Orthodontic GCF | Baseline, 1hour, 1day, 7days, 14days, 21days and 28days
  To evaluate the amount of protein content in GCF of orthodontic patients at different force magnitudes.

OTHER OUTCOMES:
Pre-Study Bone Assessment | Before actual enrolment.
  To evaluate the amount of bone density (Hounsfield Unit, HU) around the experimental teeth in CBCT.
Pre-Study Root Length Assessment | Before actual enrolment.
  To evaluate the root length (mm) of the experimental teeth in CBCT.
Pre-Study Root Shape Assessment | Before actual enrolment.
  To evaluate the root shape (Curved or Straight) of the experimental teeth by using CBCT.
Pre-Study Root Resorption Assessment | Before actual enrolment.
  To evaluate the existence of previous apical root resorption (scoring index by Malmgren < Grade 1) of the experimental teeth by using CBCT.
Oral Health Assessment | Baseline, 1hour, 1day, 7days, 14days, 21days and 28days
  Plaque Index (PI) was monitored by using modified Silness and Löe Index.
Oral Health Assessment | Baseline, 1hour, 1day, 7days, 14days, 21days and 28days
  Gingival Index was monitored by using modified Silness and Löe Index.

CONTACTS AND LOCATIONS:
Overall Officials: Harraa S. Mohammed-Salih, MSc., Principal Investigator — University of Baghdad
Locations (1):
- Harraa Sabah Mohammed-Salih, Baghdad, Iraq

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Saloom HF, Papageorgiou SN, Carpenter GH, Cobourne MT. Impact of Obesity on Orthodontic Tooth Movement in Adolescents: A Prospective Clinical Cohort Study. J Dent Res. 2017 May;96(5):547-554. doi: 10.1177/0022034516688448. Epub 2017 Jan 23. PMID 28113000
- [Background] Rody WJ Jr, Holliday LS, McHugh KP, Wallet SM, Spicer V, Krokhin O. Mass spectrometry analysis of gingival crevicular fluid in the presence of external root resorption. Am J Orthod Dentofacial Orthop. 2014 Jun;145(6):787-98. doi: 10.1016/j.ajodo.2014.03.013. PMID 24880850
- See also: Orthodontic Root Resorption — https://medlineplus.gov/